CLINICAL TRIAL: NCT00054574
Title: A Clinical Trial Evaluating The Safety And Efficacy Of ABX-EGF In Patients With Hormone Resistant Prostate Cancer With Elevated PSA Without Metastasis
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269889; UCLA-0206074; ABX-0301
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: panitumumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as ABX-EGF can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of ABX-EGF in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical effect of monoclonal antibody ABX-EGF, determined by the PSA response, in patients with hormone-resistant prostate cancer with rising PSA values without metastasis.
* Determine the pharmacokinetics and safety profile (including immunogenicity) of this drug in these patients.
* Determine the overall survival of patients treated with this drug.
* Determine the time to disease progression and time to PSA progression in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive monoclonal antibody ABX-EGF IV over 1 hour once weekly. Treatment continues every 8 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: Approximately 30-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer with rising PSA values without metastasis

  * PSA must be at least 5 ng/mL
  * PSA must show an increase above a reference level on 2 separate occasions
* Must have tumor over-expressing epidermal growth factor receptor (EGFr) by immunohistochemistry

  * Staining must be 2+ or 3+ in at least 10% of evaluated tumor cells
  * Must have tissue available for diagnostics
* Must have failed prior front-line luteinizing hormone-releasing hormone (LHRH) analogue (e.g., leuprolide or goserelin) OR failed orchiectomy and have castrate levels of testosterone (less than 50 mg/mL) NOTE: Must continue on a LHRH analogue (unless an orchiectomy was performed) throughout the study

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* AST and ALT no greater than 3 times ULN

Renal

* Creatinine less then 2.2 mg/dL
* Calcium no greater than ULN

Cardiovascular

* Left ventricular ejection fraction at least 45% by MUGA
* No myocardial infarction within the past year

Other

* HIV negative
* Fertile patients must use effective contraception during and for 1 month after study
* No other malignancy within the past 5 years except basal cell carcinoma
* No history of chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation, administration, or interpretation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics
* At least 6 weeks since prior steroidal or nonsteroidal antiandrogens (4 weeks for flutamide)
* Concurrent steroid therapy allowed as replacement therapy only

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* At least 30 days since prior investigational therapy
* At least 30 days since prior anticancer therapy
* No prior systemic therapy for prostate cancer (except hormonal therapy)
* No prior anti-EGFr therapy
* Concurrent antihypercalcemic treatment allowed in the presence of elevated calcium levels but not as cancer therapy for bone disease
* No other concurrent anti-EGFr therapy
* No other concurrent anticancer therapy
* No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2003-09 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Belldegrun, MD, FACS, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania